CLINICAL TRIAL: NCT07343258
Title: Pilot Study on Follow-Up of (Acutely) Suicidal Individuals From the Flemish Suicide Helpline, Zelfmoordlijn 1813, to Promote Continuity of Care
Brief Title: Pilot Study on Follow-Up of (Acutely) Suicidal Individuals From the Flemish Suicide Helpline
Acronym: CONT-1813
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ONZ-2025-0344
Record Dates: First submitted 2025-11-26; First posted 2026-01-15 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Suicide; Suicidal Ideation and Behavior; Crisis Intervention
Keywords: suicidal ideation; suicide-related coping; suicidal behavior; crisis line
MeSH Terms: conditions — Suicide; Suicidal Ideation; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Callers, responders and callback callers involved in callback conversations at Suicide Line 1813 (Experimental): The main target group of this research are (acutely) suicidal individuals who contact Zelfmoordlijn 1813 by phone and consent to receive callback conversations followed by an interview to share their experiences.
  During the pilot study, a number of experienced call responders (i.e., trained volunteers of the Zelfmoordlijn 1813 who offer callers a callback trajectory) and callback callers (i.e., staff members of the CPZ who conduct the callback conversations) apply the callback methodology developed by the CPZ. Call responders and callback callers will also be interviewed to provide further insights into the callback methodology.
  Interventions: Other: Callbacks from the Zelfmoordlijn 1813

INTERVENTIONS:
Other: Callbacks from the Zelfmoordlijn 1813 — Callers of Zelfmoordlijn 1813 are called back after their initial conversation, in which they themselves contacted the Zelfmoordlijn 1813. The callbacks focus on crisis management at the Zelfmoordlijn 1813 and are not intended as a form of formal support. During the callback calls, the specific needs of the caller are addressed, tailored to the callback profile assigned by a call responder based on the initial call. There are three different callback profiles for callers: (1) those for whom the crisis call immediately focuses on creating safety, with the callback calls further reinforcing this safety, (2) those for whom the focus is on crisis management, with follow-up aimed at developing and implementing a Safety Plan, and (3) those who experience barriers to discussing their suicidal thoughts, with the callback conversations being used to facilitate the step towards professional help or to make suicide discussable within their own network or existing support services.

SUMMARY:
This pilot study aims to assess the acceptance, feasibility, and added value of follow-up calls at the suicide helpline, Zelfmoordlijn 1813, in Flanders (Belgium). It serves as a crucial preparatory step in the development and implementation process of the callback methodology at Zelfmoordlijn 1813.

DETAILED DESCRIPTION:
International research confirms the importance of suicide prevention helplines. They offer immediate crisis support and try to guide people toward appropriate assistance. In practice, however, many callers do not follow up on referrals. Barriers such as costs, waiting times, or insufficient motivation play a role in this. Although call responders mainly offer emotional support, one conversation is often not enough to go into depth on concrete strategies or referrals. Nevertheless, in addition to offering a listening ear, helplines can play a crucial role in motivating and activating callers to seek further help.

The effectiveness of an initial crisis intervention is strongly related to the extent to which it is embedded in a broader care process. That is why there is growing international attention for systematic follow-up after an initial call to a helpline. International studies convincingly show that follow-up conversations after a crisis call have positive effects. Follow-up calls offer extra support, help people take the step towards (professional) help, and reinforce self-care strategies. In the United States, such calls were funded and organized by the health service SAMHSA. In Ireland, research showed that people who were called back after an initial call were significantly less likely to die by suicide than people who did not receive follow-up. In a large-scale American study, nearly 80% of suicidal callers said that the follow-up calls had helped them prevent suicide. More than 90% felt safer afterwards. People at acute risk of suicide in particular reported benefiting from the calls, which they found motivating and protective. Multiple and longer follow-up calls were associated with a stronger sense of safety and a lower estimated risk of suicide. Elements such as safety planning and strengthening social support proved to be decisive in this regard.

In this context, the Flemish Expertise Center for Suicide Prevention (VLESP, Ghent University), in collaboration with the Center for Suicide Prevention (CPZ), is investigating whether and how telephone follow-up calls are feasible for adult callers to the Zelfmoordlijn 1813 who are at (acute) risk of suicide. This is an exploratory pilot study that examines whether this form of follow-up is practically feasible and what added value it can offer as a supplement to the existing services. In this pilot study, CPZ staff members, known as callback callers, conduct callback conversations with a limited group of callers who have previously contacted the Zelfmoordlijn 1813 and given their consent to be called back for research purposes. The callback method provides for a maximum of three callback conversations per person, each of which responds to the individual needs of the caller. The callback method distinguishes between three callback profiles: safety conversation, safety planning, and continuity of care.

During this pilot study, callers are recruited with the help of a limited group of experienced volunteers from the Zelfmoordlijn 1813. These volunteers remain anonymous to the outside world and play a central role in the recruitment process. During the telephone conversation, they assess whether the caller meets the selection criteria for participation in the callback study. If the caller is 18 years of age or older, is calling from a personal telephone, and could benefit from a callback, the caller is invited to participate in the study.

Qualitative interviews with both callers and callback callers and focus groups with call responders are used to assess how the callback method is perceived. Aspects such as acceptance, feasibility, and perceived added value are examined. The interviews with callers and callback callers each last approximately one hour. Conversations with callers take place by telephone, while interviews with callback callers are conducted at the CPZ office. The focus groups with call responders last approximately two hours. Responders can choose to participate in an online session or a physical meeting at the CPZ office. A total of between 53 and 98 persons will participate in the study, namely: 3 callback callers from the CPZ, 20 call responders from the Zelfmoordlijn 1813, and between 30 and 75 participating callers.

The findings from this pilot study will serve as a basis for further refining the callback methodology at Zelfmoordlijn 1813 and, if regarded as positive, preparing for broader implementation.

ELIGIBILITY:
1. Callers

   Inclusion criteria:
   * The caller is 18 years or older.
   * The caller speaks Dutch.
   * The caller calls the Zelfmoordlijn 1813 for themselves due to suicidal ideation.
   * The caller must benefit from callback conversations fitting one of the three callback profiles.
   * The caller is not a frequent caller to the Zelfmoordlijn 1813.
   * The caller can be called back directly on a personal device.
   * The caller is legally competent, meaning they can oversee the potential consequences of participation, such as time investment and availability.
   * At the time of recruitment, the caller is not receiving support within a care trajectory where attention is paid to their suicidality. Or the care provider is not available quickly enough (e.g., due to maternity leave) if the caller falls within the callback profile focusing on a safety conversation.

   Exclusion criteria:
   * The caller is younger than 18 years.
   * The caller does not speak Dutch.
   * The caller does not call the Zelfmoordlijn 1813 for themselves.
   * The caller is a frequent caller to the Zelfmoordlijn 1813.
   * The call responder assesses that urgent medical help is necessary.
   * The caller expresses a homocide threat during the original conversation to the Zelfmoordlijn 1813.
   * The caller cannot be called back on a personal device (e.g., persons in detention).
   * The caller is not legally competent to oversee the consequences of participation (e.g., under the influence of alcohol and/or drugs).
   * At the time of recruitment, the caller is receiving support within a care trajectory where attention is paid to their suicidality.
2. Call responders The CPZ chooses to recruit call responders who have extensive experience in answering calls at the Zelfmoordlijn 1813. Therefore, not all call responders of the Zelfmoordlijn 1813 are trained to recruit callers.
3. Callback callers The staff members of the CPZ who are involved in developing and implementing the callback methodology will also participate in the research by means of an interview.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Experiences of callers, responders and callback callers with the callback methodology from the Zelfmoordlijn 1813 | Participating callers will be interviewed 7 to 14 days after completing their callback trajectory, callback callers within 2 to 3 weeks after the final callback of the study and call responders within 1 month after completing recruitment.
  Qualitative data is collected through semi-structured telephone interviews with callers who participated in the callback trajectory, each lasting approximately one hour. To examine the callback methodology of Zelfmoordlijn 1813 from the perspective of callers, interview guidelines were developed aiming to gain insight into the acceptance, feasibility, added value and barriers of the callback conversations. In addition to the caller interviews, the experiences of call responders in recruiting callers for follow-up are captured during focus group discussions. The experiences of callback callers with implementing the callback methodology are equally mapped during semi-structured interviews.

OTHER OUTCOMES:
Socio-demographic variables of callers | At the moment of enrollment
  Gender and age

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Portzky, PhD, Principal Investigator — University Ghent
Locations (1):
- Flemish Centre of Expertise in Suicide Prevention, Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No